CLINICAL TRIAL: NCT03900715
Title: A Phase 2, Multicenter, Single-arm Study to Evaluate the Efficacy, Pharmacokinetics, and Safety of Luspatercept (ACE-536) for the Treatment of Anemia Due to IPSS-R Very Low, Low or Intermediate Risk Myelodysplastic Syndromes (MDS) in Japanese Subjects Who Are Not Requiring Red Blood Cell Transfusion
Brief Title: An Efficacy and Safety Study of Luspatercept (ACE-536) for the Treatment of Anemia Due to IPSS-R Very Low, Low or Intermediate Risk Myelodysplastic Syndromes (MDS) in Japanese Subjects Who Are Not Requiring Red Blood Cell Transfusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-536-MDS-003; U1111-1224-6268 (Registry Identifier: WHO)
Record Dates: First submitted 2019-03-14; First posted 2019-04-03 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; MDS; ACE-536; Anemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luspatercept Administration (Experimental): Luspatercept will be administered as a subcutaneous injection every 3 week (21 days; Q3W), at an initial dose level of 1.0 mg/kg. Doses may be titrated up starting at dosing visit Week 7 Day 1 (W7D1)
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Luspatercept

SUMMARY:
The study will be conducted in compliance with the International Council for Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

This is a Phase 2, multicenter, single-arm study to evaluate the efficacy, safety and Pharmacokinetics (PK) of luspatercept (ACE-536) for the treatment of anemia due to International prognostic scoring system-Revised (IPSS-R) very low, low or intermediate risk Myelodysplastic syndromes (MDS)in Japanese subjects who are not requiring Red blood cell (RBC) transfusion.

The study is divided into the Screening Period, a Treatment Period and a Post-Treatment Follow up Period.

DETAILED DESCRIPTION:
Anemia is considered to be one of the most prevalent cytopenias in patients who have myelodysplastic syndromes, an umbrella term used to describe disorders relating to the ineffective production of red blood cells, white blood cells, and/or platelets. Ranging in severity from mild (asymptomatic) to severe, anemia can result in patients requiring regular red blood cell (RBC) transfusions, which can lead to further complications from iron overload. The goal of this study is to assess the efficacy, safety and PK of luspatercept in anemic patients who are categorized as International Prognostic Scoring System-Revised (IPSS-R) very low, low, or intermediate risk Myelodysplastic syndrome (MDS), and not requiring RBC transfusion. Subjects deemed eligible for the study will be enrolled and treated with luspatercept. Best supportive care (BSC) may be used in combination with study treatment when clinically indicated per investigator. Best supportive care includes, but is not limited to, treatment with transfusions, antibiotic, antiviral and/or antifungal therapy, and nutritional support as needed. Best supportive care for this study excludes the use of ESAs. Patients should receive treatment up to a minimum of 24 weeks after which an MDS Disease assessment visit is scheduled to assess the response to treatment. Patients who are determined to be experiencing clinical benefit may continue treatment. Continued clinical benefit will be re-assessed every 24 weeks. Once patients are discontinued from study treatment, they will enter a post treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 20 years of age the time of signing the informed consent form (ICF)
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject has a documented diagnosis of MDS according to WHO 2016 classification that meets IPSS-R classification of very low, low, or intermediate risk disease, and:

   • < 5% blasts in bone marrow
5. Subject has symptomatic anemia with mean Hgb concentration < 10.0 g/dL from 2 measurements (one performed within 1 day prior to W1D1 and the other performed 7 to 35 days prior to W1D1) that does not require RBC transfusion. If more than one measurement exists in the period of 7 to 35 days prior to W1D1, the most recent value will be used.
6. Subject must be TI, as documented by the following criteria:

   • No RBC transfusion administered within 16 weeks prior to W1D1 (except transfusions due to blood loss or infection that occurred between 16 and 8 weeks prior to W1D1)
7. Subject has Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2
8. Females of childbearing potential (FCBP), defined as a sexually mature woman who:

1) has achieved menarche at some point, 2) not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy or amenorrhea due to other medical reasons does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months), must:

* Have two negative pregnancy tests as verified by the investigator prior to starting study therapy (unless the screening pregnancy test was done within 72 hours of W1D1). She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence1 from heterosexual contact.
* Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, highly effective contraception without interruption, 5 weeks prior to starting investigational product, during the study therapy (including dose interruptions), and for 12 weeks after discontinuation of study therapy.
* If breastfeeding, agree to stop breastfeeding prior to the participation in the study and not to resume breastfeeding after treatment discontinuation.

  9. Male subjects must:
* Practice true abstinence2 (which must be reviewed prior to each IP administration or on a monthly basis [eg, in the event of dose delays]) or agree to use a condom (latex or non-latex, but not made out of natural [animal] membrane) during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 12 weeks following investigational product discontinuation, even if he has undergone a successful vasectomy.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject with the any of the following prior treatments for underlying disease:

   * Disease modifying agents (eg, immune-modulatory drug [IMiDs such as lenalidomide])

     - Except if the subject received ≤ 1 week of treatment with a disease modifying agent ≥ 8 weeks from W1D1, at the investigator's discretion.
   * Hypomethylating agents

     - Subjects may be enrolled at the investigator's discretion contingent that the subject received no more than 2 injections of HMA. The last dose must be ≥ 8 weeks from the date of W1D1.
   * Luspatercept (ACE-536) or sotatercept (ACE-011)
   * Allogeneic and/or autologous hematopoietic cell transplant
2. Subject with myelodysplastic syndromes/myeloproliferative neoplasms (MDS/MPN) according to WHO 2016 classification (ie, chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (aCML), BCR-ABL12, juvenile myelomonocytic leukemia (JMML), MDS/MPN unclassifiable.
3. Subject with secondary MDS, ie, MDS that is known to have arisen as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases.
4. Subject with known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or hypothyroidism, or any type of known clinically significant bleeding or sequestration. Subject with drug induced anemia (eg, mycophenolate).

   • Iron deficiency to be determined by serum ferritin < 100 μg/L and additional testing if clinically indicated (eg, calculated transferrin saturation [iron/total iron binding capacity ≤ 20%] or bone marrow aspirate stain for iron).
5. Subject with known history of diagnosis of AML
6. Subject receiving any of the following treatment within 8 weeks prior to W1D1:

   * Anticancer cytotoxic chemotherapeutic agent or treatment
   * ESAs
   * Granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colonystimulating factor (GM-CSF), unless given for treatment of febrile neutropenia
   * Immunosuppressive therapy for MDS
   * Systemic corticosteroid, except for subjects on a stable or decreasing dose for ≥ 1 week prior to W1D1 for medical conditions other than MDS
   * Other RBC hematopoietic growth factors (eg, Interleukin-3)
   * Androgens, unless to treat hypogonadism
   * Hydroxyurea, anagrelide
   * Oral retinoids
   * Arsenic trioxide
   * Interferon and interleukins
   * Investigational drug or device, or approved therapy for investigational use (if 5 times the half-life of the previous investigational drug exceeds 8 weeks, then the time of exclusion should be extended up to 5 times the half-life of the investigational drug)
7. Subject with uncontrolled hypertension, defined as repeated elevations of systolic blood pressure (SBP) of ≥ 150 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg despite adequate treatment, or with a history of hypertensive crisis or hypertensive encephalopathy.
8. Subject with any of the following laboratory abnormalities:

   * Absolute neutrophil count (ANC) < 500/μL (0.5 x 10^9/L)
   * Platelet count < 30,000/μL (30 x 10^9/L) (Exclude subjects that may be at risk of bleeding regardless of platelet counts. This includes [but is not limited to] subjects currently using aspirin or heparin, immediately after surgery, or easily causes bleeding such as nasal bleeding or subcutaneous bleeding or previous episode of major bleeding where the cause was not effectively treated.)
   * Estimated glomerular filtration rate (eGFR) < 40 mL/min/1.73 m^2 (via the 4-variable modification of diet in renal disease [MDRD] formula, Appendix G)
   * Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) or alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT) ≥ 3.0 x upper limit of normal (ULN)
   * Total bilirubin ≥ 2.0 x ULN. - Higher levels are acceptable if these can be attributed to active red blood cell precursor destruction within the bone marrow (ie, ineffective erythropoiesis) or in the presence of known history of Gilbert Syndrome.
9. Subject with prior history of malignancies, other than MDS, unless the subject has been free of the disease for ≥ 5 years. However, subjects with the following history/concurrent conditions are allowed if considered as curatively treated:

   * Basal or squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system)
10. Subject with major surgery within 8 weeks prior to W1D1. Subjects must have completely recovered from any previous surgery prior to W1D1
11. Subject with history of cerebrovascular accident (including ischemic, embolic, and hemorrhagic cerebrovascular accident), transient ischemic attack, deep venous thrombosis (DVT; including proximal and distal), pulmonary or arterial embolism, arterial thrombosis or other venous thrombosis within 6 months prior to W1D1 Note: prior superficial thrombophlebitis is not an exclusion criterion.
12. Subject with the following cardiac conditions within 6 months prior to W1D1:

    myocardial infarction, uncontrolled angina, acute decompensated cardiac failure or New York Heart Association (NYHA) Class III-IV heart failure, or uncontrolled cardiac arrhythmia as determined by the investigator. Subjects with a known ejection fraction ˂35%, confirmed by a local echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan performed within 6 months prior to W1D1.
13. Subject with uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment).
14. Subject with known human immunodeficiency virus (HIV), known evidence of active infectious hepatitis B, and/or known evidence of active Hepatitis C. Local laboratory testing confirming HIV, hepatitis B, and hepatitis C status should not have been performed beyond 4 weeks prior to the date of ICF signature.
15. Subject with history of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in luspatercept (see current IB).
16. Pregnant or breastfeeding females.
17. Subject has any significant medical condition, laboratory abnormality, psychiatric illness, or is considered vulnerable by local regulations (eg, imprisoned or institutionalized) that would prevent the subject from participating in the study.
18. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
19. Subject has any condition or receives concomitant medication that confounds the ability to interpret data from the study.
20. Subject has history of active SARS-CoV-2 infection within 4 weeks prior to screening, unless the subject has adequately recovered from COVID-19 symptoms and related complications as per investigator's discretion and following a discussion with the Medical Monitor. Use of a live COVID-19 vaccine is prohibited within 4 weeks prior to W1D1.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- Japan (19):
  - Local Institution - 338, Matsuyama, Ehime
  - Local Institution - 344, Nagasaki, Nagasaki
  - Local Institution - 336, Sayama, Osaka
  - Local Institution - 345, Chiba
  - Local Institution - 334, Fukuoka
  - Local Institution - 347, Himeji
  - Local Institution - 337, Hitachi, Ibaraki
  - Local Institution - 346, Kamakura
  - Local Institution - 331, Kamogawa
  - Local Institution - 348, Kitakyushu
  - Local Institution - 349, Kofu
  - Local Institution - 343, Nagoya
  - Local Institution - 335, Okayama
  - Local Institution - 342, Osaka
  - Local Institution - 341, Ōgaki
  - Local Institution - 333, Sagamihara
  - Local Institution - 339, Sendai
  - Local Institution - 332, Shibuya-ku
  - Local Institution - 330, Shinagawa-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Luspatercept: Participants are administered luspatercept (ACE-536): starting dose of 1.0 mg/kg subcutaneous injection every 3 weeks (21 days; Q3W).
Period: Overall Study
Arm/Group | Luspatercept
Started | 21
Efficacy Evaluable Population (Participants who received at least one dose of luspatercept and had at least two hemoglobin assessments ≥ 8 weeks apart post-treatment.) | 19
Completed | 0
Not Completed | 21
Not completed — Protocol Deviation | 1
Not completed — Lack of Efficacy | 1
Not completed — Progressive Disease | 6
Not completed — Adverse Event | 2
Not completed — Other reasons | 11

BASELINE CHARACTERISTICS:
Arm/Group | Luspatercept
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.5 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Asian (Japanese) | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Not Hispanic or Latino | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Hematologic Improvement in Erythroid Response (HI-E) Per International Working Group (IWG) Through Week 24
Description: Hematologic improvement is defined as the percent of participants meeting HI-E criteria of >= 1.5 g/dL increase in hemoglobin (Hgb) sustained over any consecutive 56-day period in the absence of red blood cell (RBC) transfusions from Week 1 Day 1 through Week 24. Participants who discontinued from the Treatment Period without achieving HI-E are counted as non-responders.
Time Frame: Week 1 Day 1 through Week 24
Population: Intent-to-Treat Population: All enrolled participants regardless of whether or not the participant received luspatercept.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept
Number analyzed (Participants) | 21
Percentage of participants | 47.6 [25.7 to 70.2]

2. Secondary Outcome: Percentage of Participants Who Achieved Modified Hematologic Improvement in Erythroid Response (mHI-E) Per International Working Group (IWG)
Description: Modified hematologic improvement is defined as the percent of participants meeting mHI-E criteria of >= 1.5 g/dL mean increase in hemoglobin (Hgb) compared to baseline sustained over any consecutive 56-day period in the absence of red blood cell (RBC) transfusions from Week 1 Day 1 through Week 24 and Week 48 of the Treatment Period. Participants who discontinued from the Treatment Period without achieving mHI-E are counted as non-responders. Baseline Hgb is defined as the mean of the two central laboratory values (one performed within 1 day prior to W1D1 and the other performed 7 to 35 days prior to W1D1).
Time Frame: Week 1 Day 1 through Week 24 and Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept
Number analyzed (Participants) | 21
Percentage of participants
  Week 1 Day 1 through Week 24 | 57.1 [34.0 to 78.2]
  Week 1 Day 1 through Week 48 | 66.7 [43.0 to 85.4]

3. Secondary Outcome: Percentage of Participants Who Achieved Hematologic Improvement in Erythroid Response (HI-E) Per International Working Group (IWG) Through Week 48
Description: Hematologic improvement is defined as the percent of participants meeting HI-E criteria of >= 1.5 g/dL increase in hemoglobin (Hgb) sustained over any consecutive 56-day period in the absence of red blood cell (RBC) transfusions from Week 1 Day 1 through Week 48 of the Treatment Period. Participants who discontinued from the Treatment Period without achieving HI-E are counted as non-responders.
Time Frame: Week 1 Day 1 through Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept
Number analyzed (Participants) | 21
Percentage of participants | 57.1 [34.0 to 78.2]

4. Secondary Outcome: Time to Hematologic Improvement in Erythroid Response (HI-E)
Description: Defined as time from Week 1 Day 1 to first onset of achieving ≥ 1.5 g/dL increase in hemoglobin (Hgb) over any consecutive 56-day period in the absence of red blood cell (RBC) transfusions.
Time Frame: Week 1 Day 1 through Week 24 and Week 48
Population: All treated participants who achieve HI-E until week 24 and 48.
Measure: Median (Full Range); unit: Days
Arm/Group | Luspatercept
Number analyzed (Participants) | 12
Days
  Week 1 Day 1 through Week 24: number analyzed (Participants) | 10
  Week 1 Day 1 through Week 24 | 26.5 [14 to 87]
  Week 1 Day 1 through Week 48 | 36.5 [14 to 275]

5. Secondary Outcome: Time to Modified Hematologic Improvement in Erythroid Response (mHI-E)
Description: Defined as the time from Week 1 Day 1 to first onset of achieving ≥ 1.5 g/dL mean increase in hemoglobin (Hgb) compared to baseline over any consecutive 56-day period in the absence of red blood cell (RBC) transfusions. Baseline Hgb is defined as the mean of the two central laboratory values (one performed within 1 day prior to W1D1 and the other performed 7 to 35 days prior to W1D1.
Time Frame: Week 1 Day 1 through Week 24 and Week 48
Population: All treated participants who achieve mHI-E until week 24 and 48.
Measure: Median (Full Range); unit: Days
Arm/Group | Luspatercept
Number analyzed (Participants) | 14
Days
  Week 1 Day 1 through Week 24: number analyzed (Participants) | 12
  Week 1 Day 1 through Week 24 | 0.0 [0 to 8]
  Week 1 Day 1 through Week 48 | 0.0 [0 to 210]

6. Secondary Outcome: Duration of Hematologic Improvement in Erythroid Response (HI-E)
Description: Defined as the maximum duration of achieving ≥ 1.5 g/dL increase in hemoglobin (Hgb) for participants who achieve Hgb increase ≥ 56 days in the absence of red blood cell (RBC) transfusions. Participants who maintain HI-E through the end of the Treatment Period or time of analysis will be censored at the date of treatment discontinuation/time of analysis or death, whichever occurs first.
Time Frame: Week 1 Day 1 through end of treatment period (up to an average of 74 weeks and maximum of 178 weeks)
Population: All treated participants who achieve HI-E
Measure: Median (Full Range); unit: Weeks
Arm/Group | Luspatercept
Number analyzed (Participants) | 13
Weeks | 40.0 [30.1 to 57.9]

7. Secondary Outcome: Duration of Modified Hematologic Improvement in Erythroid Response (mHI-E)
Description: Defined as the maximum duration of achieving ≥ 1.5 g/dL increase in hemoglobin for participants who achieve mean hemoglobin (Hgb) increase compared to baseline ≥ 56 days in the absence of red blood cell (RBC) transfusions. Participants who maintain mHI-E through the end of the Treatment Period or time of analysis will be censored at the date of treatment discontinuation/time of analysis or death, whichever occurs first. Baseline Hgb is defined as the mean of the two central laboratory values (one performed within 1 day prior to W1D1 and the other performed 7 to 35 days prior to W1D1.
Time Frame: Week 1 Day 1 through end of treatment period (up to an average of 74 weeks and maximum of 178 weeks)
Population: All treated participants who achieve mHI-E
Measure: Median (Full Range); unit: Weeks
Arm/Group | Luspatercept
Number analyzed (Participants) | 14
Weeks | 92.1 [46.1 to 157.4]

8. Secondary Outcome: Red Blood Cell Transfusion Independence (RBC-TI)
Description: Defined as the percentage of participants not being given any red blood cell (RBC) transfusion during the treatment period.
Time Frame: Week 1 Day 1 through Week 24, Week 48, and Week 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept
Number analyzed (Participants) | 21
Percentage of participants
  Week 1 Day 1 through Week 24 | 81.0 [58.1 to 94.6]
  Week 1 Day 1 through Week 48 | 81.0 [58.1 to 94.6]
  Week 1 Day 1 through Week 72 | 81.0 [58.1 to 94.6]

9. Secondary Outcome: Progression to Acute Myeloid Leukemia (AML)
Description: Number of participants progressing to acute myeloid leukemia (AML). AML progression is defined per WHO classification of ≥ 20% blasts in peripheral blood or bone marrow. Subjects with diagnosis of AML will be considered to have had an event. Subjects who have not progressed to AML at the time of analysis will be censored at the last assessment date which does not indicate progression to AML.
Time Frame: From Week 1 Day 1 up to approximately 44 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept
Number analyzed (Participants) | 21
Participants | 0

10. Secondary Outcome: Time to Acute Myeloid Leukemia (AML) Progression
Description: Defined as the time between W1D1 and first diagnosis of AML as per WHO classification of ≥ 20% blasts in peripheral blood or bone marrow. Participants with diagnosis of AML will be considered to have had an event. Participants who have not progressed to AML at the time of analysis will be censored at the last assessment date which does not indicate progression to AML.
Time Frame: Week 1 Day 1 to first diagnosis of AML (up to approximately 44 months)
Population: All treated participants with AML progression. (No participants had AML progression)
Arm/Group | Luspatercept
Number analyzed (Participants) | 0

11. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as time from Week 1 Day 1 to a participants death date or last known alive date. Participants who die, regardless of the cause of death, will be considered to have had an event. Participants who are alive at the time of analysis will be censored at the last assessment date at which the participant was known to be alive. All participants who were lost to follow-up will also be censored at the time of last contact.
Time Frame: Week 1 Day 1 to to a participants death date or last known alive date (up to approximately 44 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Luspatercept
Number analyzed (Participants) | 21
Months | NA [NA to NA] — Insufficient number of participants with events

12. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Treatment-emergent adverse events include adverse events that started on or after the first dose until 42 days after the last dose, as well as those SAEs made known to the investigator at any time thereafter that are suspected of being related to study drug. An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study.
  Grade 3 = Severe Grade 4 = Life-threatening Grade 5 = Death
Time Frame: From first dose to 42 days after last dose (up to approximately 42.5 months)
Population: Safety Population: All participants who were enrolled and received at least one dose of luspatercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept
Number analyzed (Participants) | 21
Participants
  Treatment-Emergent Adverse Events (TEAEs) | 20
  Suspected Drug Related TEAE | 8
  Serious TEAE | 6
  Suspected Drug Related Serious TEAE | 1
  Grade 3 or 4 TEAE | 8
  Suspected Drug Related Grade 3 or 4 TEAE | 4
  Grade 5 TEAE | 0
  Suspected Drug Related Grade 5 TEAE | 0
  TEAE Leading to Dose Interruption | 5
  TEAE Leading to Dose Reduction | 2
  TEAE Leading to Dose Withdrawn | 6

13. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: W1D1 (pre-dose), W1D3, W2D1, W2D3, W3D1, W4D1, W10D1, W13D1, W16D1, W17D1, W18D1, W19D1, W22D1, 24-Week MDS Disease Assessment, and every 12 weeks from the 24-Week MDS Disease Assessment Visit for up to 1 year from the first dose.
Population: All participants who received at least 1 dose of luspatercept and had sufficient PK samples collected for non-compartmental analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Luspatercept
Number analyzed (Participants) | 9
ug/mL | 5.713 (29.27)

14. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Median (Full Range); unit: Day
Arm/Group | Luspatercept
Number analyzed (Participants) | 9
Day | 7.921 [2.884 to 13.75]

15. Secondary Outcome: Area Under the Concentration-Time Curve (AUC21d)
Time Frame: W1D1 (pre-dose), W1D3, W2D1, W2D3 , W3D1, W4D1 (21 days after dose administration)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*ug/mL
Arm/Group | Luspatercept
Number analyzed (Participants) | 9
Day*ug/mL | 94.28 (29.31)

16. Secondary Outcome: Number of Participants With a Positive Anti-Drug Antibody (ADA) Test
Description: Number of participants under each ADA positive category. A participant is counted as 'Treatment-Emergent' if there is a positive post-baseline sample while the baseline sample is ADA negative, or there is a positive post-baseline sample with a titer >= 4-fold of the baseline titer while the baseline sample is ADA positive. A participant is counted as 'Preexisting' if the baseline sample is ADA positive and the participant is not qualified for 'Treatment-Emergent'. Positive to preexisting ADA is considered baseline sample is positive and all post-baseline samples are negative, or both baseline and post-baseline samples are positive, but all positive post-baseline sample have a titer < 4-fold of the baseline titer.
Time Frame: W1D1 (must be collected before the first dose), W4D1, W10D1, W16D1, W22D1, 24-Week MDS Disease Assessment Visit and every 12 weeks (± 14 days) from the 24-Week MDS Disease Assessment Visit for up to 1 year from the first dose..
Population: Safety Population: all participants who were enrolled and received at least one dose of luspatercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept
Number analyzed (Participants) | 21
Participants
  Preexisting | 0
  Treatment-Emergent | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose until their study completion (up to approximately 44 months). SAEs and other AEs were assessed from first dose to 42 days after last dose (up to approximately 42.5 months).
Arm/Group | Luspatercept
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 6/21
Other Adverse Events (participants affected / at risk) | 14/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Luspatercept (N=21)
Bronchitis (Infections and infestations) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Luspatercept (N=21)
Constipation (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Injection site pruritus (General disorders) | 2
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 2
Conjunctivitis (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 3
Blood creatinine increased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT03900715/Prot_SAP_000.pdf